CLINICAL TRIAL: NCT03479476
Title: A Double-Blind, Placebo-Controlled Trial of Metformin in Individuals With Fragile X Syndrome
Brief Title: A Trial of Metformin in Individuals With Fragile X Syndrome
Acronym: Met
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: University of Alberta (Other); St. Justine's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1068417
Record Dates: First submitted 2018-03-20; First posted 2018-03-27 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Fragile X Syndrome; Fragile X Mental Retardation Syndrome; Mental Retardation, X Linked; Genetic Diseases, X-Linked; Trinucleotide Repeat Expansion; Fra(X) Syndrome; Intellectual Disability; FXS; Neurobehavioral Manifestations; Sex Chromosome Disorders
Keywords: Congenital Abnormalities; Metformin; Nervous System Diseases; Chromosome Disorders
MeSH Terms: conditions — Fragile X Syndrome; X-Linked Intellectual Disability; Genetic Diseases, X-Linked; Intellectual Disability; Neurobehavioral Manifestations; Sex Chromosome Disorders; Congenital Abnormalities; Nervous System Diseases; Chromosome Disorders | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo Medication (Placebo Comparator): The placebo will be dosed in a weight-dependent manner. Liquid placebo will be provided to any participants unable to swallow the placebo capsules. For participants under 50kg at baseline, the initial dose will be 250mg once per day, and if this dose is well tolerated, they will increase each week by 250mg until a maximum dose of 1000mg daily is reached. For participants at and above 50kg at baseline, the initial dose will be 500mg once per day, and if this dose is well tolerated, they will increase each week by 500mg until a maximum dose of 2000mg daily is reached. After the 4-week titration period, each participant will continue dosing at his or her maximum tolerated dose daily for the remaining 12 weeks of the study.
  Interventions: Drug: Placebo Medication
- Active Metformin Medication (Active Comparator): The active metformin medication will be dosed in a weight-dependent manner. Liquid metformin (100mg/cc) will be provided to any participants unable to swallow the metformin capsules. For participants under 50kg at baseline, the initial dose will be 250mg once per day, and if this dose is well tolerated, they will increase each week by 250mg until a maximum dose of 1000mg daily is reached. For participants at and above 50kg at baseline, the initial dose will be 500mg once per day, and if this dose is well tolerated, they will increase each week by 500mg until a maximum dose of 2000mg daily is reached. After the 4-week titration period, each participant will continue dosing at his or her maximum tolerated dose daily for the remaining 12 weeks of the study.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Placebo Medication — Placebo liquid or capsules given in parallel to active medication.
  Other Names: Placebo
  Arms: Placebo Medication
Drug: Metformin — Active medication.
  Other Names: Glumetza; Glucophage; Fortamet; Riomet
  Arms: Active Metformin Medication

SUMMARY:
This study is a controlled trial of metformin in individuals with fragile X syndrome between the ages of 6 and 25 years. Participants will be randomized in a double-blind design to either drug or placebo and will attend three visits to the study site in a 4-month period for a series of tests. The primary objectives are to assess safety, tolerability, and efficacy of metformin in the treatment of language deficits, behavior problems, and obesity/excessive appetite in individuals with fragile X syndrome.

DETAILED DESCRIPTION:
This is a multi-site study for fragile X syndrome (FXS) patients aged 6 to 25 years inclusive. It is a randomized, double-blind, placebo-controlled trial of metformin (also known as Glumetza, Glucophage, Fortamet), a type 2 diabetes medication that can also improve obesity and excessive appetite.

Metformin has emerged as a candidate drug for the targeted treatment of FXS based on animal studies showing rescue of multiple phenotypes in the FXS model. Metformin may contribute to normalizing signaling pathways in FXS in the central nervous system, which may include activities of mTOR and PI3K, both of which have shown to be pathogenically overactive in FXS. In addition, metformin inhibits phosphodiesterase, which would lead to correction of cAMP levels, and MMP9 production, which is also elevated in FXS. Looking at the potential signaling pathways, metformin appears to be a good candidate for targeting several of the intracellular functions in neurons disrupted in FXS and, therefore, has potential to rescue several types of symptoms in individuals with FXS. The researchers have utilized metformin in the clinical treatment of over 20 individuals with FXS between the ages of 4 and 58 years and have found the medication to be well tolerated and to provide benefits not only in lowering weight gain and normalizing appetite but also in language and behavior. In this controlled trial, the researchers hope to further assess metformin's safety and benefits in the areas of language and cognition, eating and weight loss, and overall behavior.

Each participant will be involved in this trial for a period of 4 months. This will include 3 visits to the UC Davis MIND Institute and 5 phone calls. At each visit, the researchers will assess behavioral, cognitive, and language development. The researchers will also assess the side effects of the study medication throughout the trial.

Study record updated 9/26/2018 to reflect the following IRB-approved protocol modifications: Erroneous references to "digital" books for primary outcome measure were removed, as this measure is administered using print (non-digital) materials. Eligibility criteria were updated to include subjects with IQ of up to and including 79 on the Leiter-III at screening. The Hyperphagia Questionnaire (HQ-CT) was replaced by the Anxiety Depression and Mood Screen (ADAMS) as a secondary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Molecular genetic confirmation of the full FMR1 mutation or mosaicism.
* Males and non-pregnant, non-lactating females age 6 to 25 years, inclusive.
* Ability of subject and/or caregiver to understand, read, write, and speak English fluently to complete study-related materials.
* IQ ≤ 79 as measured by the Leiter-III at screening.
* Participant is able to speak at least occasional 3-word phrases.
* Participant and parent/caregiver are willing to participate in the protocol and able to attend the clinic regularly and reliably.
* Stable concomitant medication dose and dosing regimen for at least 4 weeks prior to the screening/baseline visit, and the intention to maintain a stable regimen of allowed concomitant medications for the full duration of the study.
* Stable behavioral/educational treatments for at least 4 weeks prior to the screening/baseline visit.
* Sexually active women of childbearing potential must be using a medically acceptable method of birth control for the duration of the study and have a negative urine pregnancy test collected at the initial screening/baseline visit.
* For participants who are not their own legal guardian, the parent/legal authorized representative is able to understand and sign an informed consent to participate in the study.

Exclusion Criteria:

* Non-cooperation or inability to follow through with the study protocol.
* Life-threatening medical problem or other major systemic illness that compromises health or safety and/or would interfere with the study.
* History of intolerable adverse events with metformin.
* Current or recent metformin treatment (within the past year).
* Body mass index (BMI) less than 2 standard deviations for age.
* Serum creatinine > 1.4 mg/dl (female) or > 1.5 mg/dl (male) at screening.
* History of metabolic acidosis or a condition with lactic acidosis.
* Severe B12 deficiency.
* Pregnancy at screening or unwillingness to use acceptable method of birth control, if applicable.

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Expressive Language Sampling (ELS) mean Number of Different Words (NDW) score | Baseline, End of Treatment/Week 16
  The ELS is collected from shared interactions around a wordless picture book involving the participant and the examiner. The primary outcome measure will be Number of Different Words (NDW) derived from transcripts of audiorecorded samples of spoken language taken from two sampling contexts (conversation and narration), according to procedures described by Abbeduto and colleagues (Abbeduto et al., 1995; Kover et al., 2012). Samples are collected pre- and post- treatment using different books on each occasion. The mean of NDW in conversation and NDW in narration will be computed, and statistically adjusted through analysis of covariance for differences in talkativeness as outlined in Conners et al., 2018. The mean NDW score ranges from 1 to infinite/unspecified. An increase (positive change) in score from baseline to follow-up indicates improvement. The greater the increase, the greater the improvement.

SECONDARY OUTCOMES:
Change from baseline in the FXS-normed Aberrant Behavior Checklist - Community Edition (ABC-C) | Baseline, Week 8, End of Treatment/Week 16
  The ABC-C is a 58-item caregiver-rated behavior scale used to examine treatment effects on challenging behaviors for individuals with FXS in the following domains: (1) irritability, agitation, crying; (2) lethargy, social withdrawal; (3) stereotypic behavior; (4) hyperactivity, noncompliance; and (5) inappropriate speech. Analysis will be performed utilizing the Sansone et al. (2012) FXS-normed ABC scoring measures.
Improvement of symptoms in FXS using the Clinical Impression - Improvement (CGI-I) scale | Baseline, Week 8, End of Treatment/Week 16
  The CGI is a clinician-rated scale utilizing history from the caregiver and incorporating it into a clinical rating, first for severity, and then for clinical follow-up. The CGI-S will be used at the baseline assessment to judge symptom severity as 1 = Normal, not at all ill; 2 = Borderline ill; 3 = Mildly ill; 4 = Moderately ill; 5 = Markedly ill; 6 = Severely ill; and 7 = Among the most extremely ill. The CGI-I will be used at the Week 8 and End of Treatment/Week 16 visits to judge the change in clinical impression as 1 = Very Much Improved; 2 = Much Improved; 3 = Minimally Improved; 4 = No Change; 5 = Minimally Worse; 6 = Much Worse; and 7 = Very Much Worse.
Change from baseline in the Visual Analog Scale (VAS) | Baseline, Week 8, End of Treatment/Week 16
  The VAS will be used to measure the severity of three specific behavioral symptoms targeted in this study: behavior problems, language abilities, and eating behavior. For each behavior the caregiver is instructed to mark their impression of the behavior at the baseline visit and again at the Week 8 and End of Treatment/Week 16 visits. The calculated distance in cm between the visit marks thereby demonstrates whether each behavior stayed the same, improved, or worsened during the study and by how much. The scale is from 0 cm (defined as "worst behavior") to 10 cm ("behavior not a problem").
Change from baseline in the Vineland Adaptive Behavior Scales-Third Edition (VABS-III) Adaptive Behavior Composite Score | Baseline, End of Treatment/Week 16
  The VABS-III is a caregiver survey interview that measures the personal and social skills of individuals from birth through adulthood. It was designed to assess handicapped and non-handicapped persons in their personal and social functioning and is appropriate for individuals of all ages. The Adaptive Behavior Composite (ABC) score is calculated from the caregiver responses using age-adjusted scoring tables. ABC scores range from 20 to 160 and indicate low (20-70), moderately low (70-85), adequate (85-115), moderately high (115-130), or high (130-160) overall adaptive functioning.
Change from baseline in the Anxiety Depression and Mood Screen (ADAMS) overall score | Baseline, Week 8, End of Treatment/Week 16
  The ADAMS consists of a series of 28 questions relating to the participant's symptoms of anxiety, depression, and mood. The sum of responses on a scale of 0 to 3 for each of the 28 questions generates the overall score, which ranges from 0 to 84. Lower scores indicate lower severity of symptoms, while higher scores indicate higher severity of symptoms. It will be completed by the caregiver at baseline, Week 8, and End of Treatment/Week 16 visits.
Change from baseline in the Child Sleep Habits Questionnaire (CSHQ) overall score | Baseline, Week 8, End of Treatment/Week 16
  The CSHQ consists of a series of questions relating to the sleep habits of children. It will be completed by caregivers of all participants, regardless of participant age, at the baseline, Week 8, and End of Treatment/Week 16 visits.
Change from baseline in the Swanson, Nolan and Pelham Questionnaire (SNAP-IV) overall score | Baseline, Week 8, End of Treatment/Week 16
  The SNAP-IV, based on DSM-V criteria for ADHD, is a caregiver-rated questionnaire that effectively identifies those with and without ADHD and accurately predicts presentation specifier (inattention, hyperactivity/impulsivity, and combined). Its psychometric properties and clinical utility have been demonstrated in multiple studies since its introduction in 2001, and it has been found to be reliable and well validated with normative data from both parents and teachers. It will be completed by caregivers of all participants at baseline, Week 8, and End of Treatment/Week 16.
Change from baseline in the Pediatric Quality of Life Questionnaire (PedsQL) Parent Proxy overall score | Baseline, Week 8, End of Treatment/Week 16
  The PedsQL Parent Proxy consists of a series of questions relating to a child's quality of life and is administered to the caregiver of the participant. The parent proxy module designed for children 8-12 years of age will be administered to the caregivers of all participants, regardless of participant age, because the questions therein are most appropriate for the overall study population's cognitive age and ability. It will be completed at the baseline, Week 8, and End of Treatment/Week 16 visits. For any participants not in school, questions pertaining to "school" will be replaced with references to "work" or other activities in their life.

CONTACTS AND LOCATIONS:
Overall Officials: Randi J Hagerman, MD, Principal Investigator — University of California, Davis
Locations (3):
- UC Davis MIND Institute, Sacramento, California, United States
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - St Justine Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/a-study-of-experimental-treatment-with-metformin-for-fragile-x-syndrome-932390/